CLINICAL TRIAL: NCT04395235
Title: Ethical Committee at Researches of Ege University
Brief Title: Perceptions of Porta Celiac Vascular Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Figen GOVSA, Prof. Dr, Senior investigator, Ege University
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: EGE18-5/45
Record Dates: First submitted 2020-04-25; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Educational Problems
Keywords: Patient-specific modelling; Graduate surgical education
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Surgical Therapy Plan (Experimental): This study pointed out that 3D surgico-anatomical models lead to more precise anatomical understanding compared to CT images in terms of detail perception. The 3D models of vascular patterns proves to be the optimal design according to the experts' evaluation with its teaching effects on surgical residents. The demonstration of the hepatic source vascular anatomy and corresponding vascular patterns may provide practically useful guides in decision making related to vascular detail during living donor liver transplantation.Model CT's were measured in order to verify 1:1 modelling and the printing the process was carried out with 3D printers of Mass Portal Pharaoh xd 20 with Eryone PLA 3D printer flament (2.2LBS)/Spool, White). Measurements of the anatomical structures were compared between the original CT images, and the CT images of the 3D model. The morphometric values such as inter-arterial distances, inter-venous distances and the distance between artery and vein were noted.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A multi-item survey was prepared to assess fellow's perception of residency training. The survey was utilized by our group, understanding of patient vascular anatomy, awareness of the changes based on variations, independent decision-making, differential diagnosis, plan on key surgical steps, and preparation for unexpected bleeding. The answers to the questions asked for each case were analyzed to include senior (3 years and over) - junior (1-2 years) residents.Assistants spend 45 minutes in the survey. Data are entered into SPSS 24.0 for statistical analysis. Wilcoxon Signed Ranks Test was used to determine any significant differences in the measurements between the original CT images, 3D rendered images, the 3D model and CT images of the 3D model. Statistical significance was defined as a p value of less than 0.05. Junior assistants stated that they perceived 2D image statistically better than 3D models compared to the senior assistants (Kruskal-Wallis Test).

SUMMARY:
Background: Primary aspect of hepatic navigation surgery is the identification of source vascular details to preserve healthy liver which has a vascularity anatomy quite challenging for the young surgeons. The purpose was to determine whether three-dimensional (3D) vascular pattern models of preoperative computed tomography images will assist resident-level trainees for hepatic surgery.

Methods: This study was based on the perception of residents who were presented with 5 different hepatic source vascular pattern and required to compare their perception level of CT, and 1:1 models in terms of importance of variability, differential of patterns and preoperative planning.

Results: All subspecialties agree that models provided better understanding of vascular source and improved preplanning. Five stations provided qualitative assessment with results showing the usefulness of porta-celiac models when used as anatomical tools in preplanning (p=0.04), simulation of interventional procedures (p=0.02), surgical education (p=0.01). None of the cases a scored less than 8.5. Responses related to understanding variations were significantly higher in the perception of the 3D model in all cases, furthermore 3D models were more useful for seniors in more complex cases 3 & 5. Some open-ended answers: "The 3D model can completely change the operation plan" One the major factors for anatomical resection of liver transplantation is the positional relationship between the hepatic arteries and the portal veins. Conclusions: The plastic-like material presenting the hepatic vascularity enables the visualization of the origin, pattern, shape, and angle of the branches with appropriate spatial perception thus making the well-structured.

DETAILED DESCRIPTION:
2.1. Research Design The study group consisted of Ege University, Faculty of Medicine general surgery residents (n:22). A five-station carousel composed of vascular patterns such as classical porta-celiac, portal vein type 2, portal vein type 3, separate branches origin of celiac trunk and portal vein pattern located between the right and the left hepatic artery. Each station contained the CT, and life size models of the cases. As data collection tool, a descriptive rating scale was used to evaluate the perceptions of each of the methods (CT and 3D solid model) in terms of their usefulness in knowing the variations, perceiving the problem, their effectiveness in differential diagnosis and preoperative planning.

Arterial variations were classified according to previous authors. In the classical anatomy, the common hepatic artery arises from the celiac trunk to form the gastroduodenal and proper hepatic arteries, and the latter dividing distally into right and left branches. Separate branches origin of the celiac trunk such as the artery from the abdominal aorta were modeled individually in cases of variant neighborhood. Portal variations were classified as the portal vein types. Type 1 is the classical appearance, in which the right portal vein and left portal are present as independent trunks. In type 2, the right anterior portal vein, right posterior portal vein, and left portal vein trifurcate from the main portal vein. In type 3, the right posterior portal vein comes directly from the middle portal vein, and the left portal vein and right anterior portal vein emerge from a common trunk.

The study was approved by the suitably constituted Ethical Committee at Researches Department of Ege University (18-5/45), within which the work was undertaken, and the study conforms to the Declaration of Helsinki. Clinicaltrails number is EGE18-6.134.

2.2. Selection of the samples The patients in this study were chosen among the ones who consulted to Ege University Faculty of Medicine, Department of General Surgery, Hepatobiliary Surgery and Transplantation Division for diagnose between September 2016 and January 2018. CT archives were screened and 100 eligible people (age: 18-62) with porta-celiac vascular patterns were selected. Patients whose radiological imaging results were suitable for modeling and the ones with no previous operation or pathology that may cause anatomical differences were included in the study.

2.3. Stations Five case carousel that could serve as an example for variational hepatic vascularity was defined with the consensus of experts in medical education, anatomy, radiology and liver transplantation team. The carousel included the following 5 cases.

Case 1. Portal vein with Type 3 classification pattern. Case 2. Normal classification porta-celiac vascular pattern. Case 3. Vascular pattern with the separate branch origin of celiac trunk. Case 4. Portal vein between the right and the left hepatic artery. Case 5. Portal vein with Type 2 classification pattern. 2.4. Image post-processing and segmentation DICOM data from CT and MRI sections of the patients were obtained using free 3D Slicer (version 4.10.1) software. Segmentations of the portal vein, hepatic vein, splenic vein were automatically generated from the venous phase, while the celiac trunk and hepatic artery were manually traced from the arterial phase.

2.5. Creating life-size patient-specific porta-celiac vascular model Model CT's were measured in order to verify 1:1 modelling and the printing the process was carried out with 3D printers of Mass Portal Pharaoh xd 20. Model production took a total of 24 hours; 4 for segmentation, 3 for editing, 15 for printing, and 1 hour for post-print processing. Arterial vessels were color-coded red, and the portal vein blue by the visualization team.

2.6. Quantitative assessment of model accuracy Measurements of the anatomical structures were performed and compared between the original CT images, and the CT images of the 3D model. The morphometric values such as inter-arterial distances (distances between arterial origins), inter-venous distances and the distance between the artery and the vein were noted. Measurements were compared for original CT images, the 3D rendered files, and the 3D vascular models. The repetition rate of the measurements which were done by two autonomous spectators, was 3 times at every scene and the mean values were taken as ultimate output and also calculated for further statistical analysis. The spectators performed with exceptional correlation (r=0.99, P<0.001).

2.7. Workshop During the workshop, 30-minute lectures were given by the expert team on variable vascular pattern, arterial structures relationship with venous structures and models in diagnosis. For each station, a period of 5-10 minutes was given.

2.8. Survey A multi-item survey was prepared to assess fellow's perception of residency training. The survey was utilized by our group, understanding of patient vascular anatomy, awareness of the changes based on variations, independent decision-making, differential diagnosis, plan on key surgical steps, and preparation for unexpected bleeding. The answers to the questions asked for each case were analyzed to include senior (3 years and over) - junior (1-2 years) residents.

2.9. Statistical analysis Data are entered into SPSS 24.0 for statistical analysis. Continuous variables were presented as mean ± standard deviation. Wilcoxon Signed Ranks Test was used to determine any significant differences in the measurements between the original CT images, 3D rendered images, the 3D model and CT images of the 3D model. Statistical significance was defined as a p value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria: General Surgery Resident -

Exclusion Criteria: General Surgery Specialist

-

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Creating life-size patient-specific porta-celiac vascular model | 05.10. 2019, 45 minutes
  The survey was utilized by our group, understanding of patient vascular anatomy, awareness of the changes based on variations, independent decision-making, differential diagnosis, plan on key surgical steps, and preparation for unexpected bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozer, Prof. Dr, Study Chair — Faculty of Medicine, Ege University; Yelda Pinar, Study Chair — Faculty of Medicine, Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The aim was to assess whether the 3D models could be more informative than the standard CT images in predicting the real cases with different patterns. We also aimed to compare the effectiveness of the life-size model with CT screen, in 5 different porta-celiac variational cases for hepatic surgery to general surgeon residents in terms of recognizing the variational vascular source, differential diagnosis and preoperative preparation stages. It also targets to evaluate the use of these models in training and proficiency exams.
Supporting Information: Study Protocol
Time Frame: Current surgical planning primarily relies on the surgeon's ability to interpret and mentally reconstruct two-dimensional (2D) CT images into 3D while planning resection margins. Although surgeons do convert what they see on flat monitors into a 3D mental design with intraoperatively expected details, each case differs from the other and 2D images are not sufficient to provide a comprehensive viewing of the vasculo-anatomical details.
Access Criteria: This will help liver transplantation team surgeons to review the most common hepatic vascular anatomy, allowing the simultaneous visualization in addition to providing the professionals with the material to be used in pedagogical curriculum.